CLINICAL TRIAL: NCT06403085
Title: THE EFFECT OF PROPRIOCEPTIVE TRAINING ON UPPER EXTREMITY FUNCTIONS AND MUSCLE ACTIVATION IN STRING INSTRUMENT PLAYERS
Brief Title: Proprioceptive Exercises in Stringed Instrument Performers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, Hasan Akbey, Firat University, Firat University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024/47
Record Dates: First submitted 2024-05-03; First posted 2024-05-07 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: String Instrument Performers
Keywords: proprioceptive education; performance; musicians

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Rhythmic Stabilization, Limb Matching, Double and Single Arm Balance, Balance with Ball and Weight Transfer will be performed for 8 weeks.
  Interventions: Other: Study group
- Control group (No Intervention): No intervention will be applied to control group

INTERVENTIONS:
Other: Study group — Rhythmic Stabilization, Limb Matching, Double and Single Arm Balance, Balance with Ball and Weight Transfer will be performed for 8 weeks.
  Arms: Study group

SUMMARY:
Musculoskeletal problems that occur in musicians are usually in the form of soft tissue injuries affecting muscles, tendons, nerves and ligaments. These injuries can cause pain, weakness and sensory changes, making it impossible to play the instrument.It is aimed to include 50 adult musicians who meet the inclusion criteria from among the performers in Elazığ Culture and Music Association, Fırat University State Conservatory Department, State Classical Turkish Music choir and musicians who are actively performing instruments within the borders of Elazığ province. Pain, posture, upper extremity function and performance will be evaluated in this study.

DETAILED DESCRIPTION:
Musculoskeletal problems that occur in musicians are usually in the form of soft tissue injuries affecting muscles, tendons, nerves and ligaments. These injuries can cause pain, weakness and sensory changes, making it impossible to play the instrument.It is aimed to include 50 adult musicians who meet the inclusion criteria from among the performers in Elazığ Culture and Music Association, Fırat University State Conservatory Department, State Classical Turkish Music choir and musicians who are actively performing instruments within the borders of Elazığ province. the aim of this study is to investigate the effects of proprioceptive training on upper extremity function and performance in musicians (stringed instrument performers). Upper Extremity Function Assessment, Upper Extremity Performance Assessment, Posture Assessment, Pain Assessment will be evaluated. Proprioceptive training will be applied 3 days a week for 8 weeks. The training will be prepared to increase the stabilization of the muscles in the shoulder, shoulder girdle and back that are active for long periods of time due to performance.

ELIGIBILITY:
Inclusion Criteria:

* Stringed instrumentalists
* Individuals between the ages of 18-65
* Musicians who have been performing for 3 years or more
* Musicians who play an instrument for at least 1 hour per day
* Musicians who want to be involved in the study as volunteers
* Musicians from whom informed consent was obtained will be included.

Exclusion Criteria:

* Upper extremity injury or surgery before the study (last 1 year)
* Individuals who are pregnant
* Individuals with psychological, neurological or systemic diseases were excluded from the study. The experimental groups of these string players will be ensured to participate regularly in the proprioceptive training protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-05-03 (Estimated); Primary Completion 2024-07-20 (Estimated); Study Completion 2024-08-20 (Estimated)

PRIMARY OUTCOMES:
Upper Extremity Performance Assessment | 10 minutes
  Purdue Pegboard test will be used for upper extremity performance evaluation. The tests will be performed with right, left and both hands. The time to complete each parameter will be recorded in seconds (sec)

SECONDARY OUTCOMES:
Upper Extremity Function Assessment | 10 minutes
  Grip and pinch strength will be assessed to evaluate upper extremity function. grip strength will be assessed using a hand dynamometer, pinch strength will be assessed using a pinchmeter

OTHER OUTCOMES:
Posture | 5 minutes
  With the DigiME device, we will evaluate the postural changes of the performers over the years due to the performance of the instrument in three dimensions (3D) and record the angular effects on the joints.
Pain Assessment | 1 minute
  Visual Analog Scale (VAS) will be used to measure the severity of pain. This scale will be numbered from 0 to 10. "0" will represent no pain and "10" will represent the highest value for perceived pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Hasan Akbey, Elâzığ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Evidence-informed physical therapy management of performance-related musculoskeletal disorders in musicians — http://pubmed.ncbi.nlm.nih.gov/25071671/